CLINICAL TRIAL: NCT01633151
Title: Validation Study for an Unobtrusive Online Sleep Measurement System
Status: Completed | Type: Observational
Sponsor: Beddit.com Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BEDDIT-2012-1
Record Dates: First submitted 2012-06-20; First posted 2012-07-04 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Apnea; Restless Legs Syndrome; Sleep Fragmentation
MeSH Terms: conditions — Apnea; Restless Legs Syndrome; Sleep Deprivation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 20 volunteers

SUMMARY:
The purpose of the study is to determine the precision of an unobtrusive sleep measurement system. The system measures a force sensor signal under the mattress and analyzes sleep quality. The system measures: time in bed, sleep stages, sleep fragmentation, heart rate, respiration rate, sleep related breathing disorders, and limb movements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Finnish-speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of 20 volunteers - 10 males, 10 females - is recruited so that their ages are distributed evenly between 18 and 80.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Precision of sleep measurement | 7 days
  The volunteers are measured for seven consecutive days. The precision of the sleep measurements output by the ubobtrusive sleep monitoring system is evaluated by comparing the measurements to polysomnography and actigraphy reference measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Markku Partinen, MD, PhD, Principal Investigator — Helsinki Sleep Clinic, Vitalmed Research Center, Helsinki, Finland
Locations (1):
- Helsinki Sleep Clinic, Vitalmed Research Centre, Helsinki, Finland